CLINICAL TRIAL: NCT01777425
Title: Long-term Control in Rhinosinusitis After FESS: Cross-sectional Observational Study on Control in Rhinosinusitis at a Mean Interval of 3 Years After FESS
Brief Title: Long-term Control in Rhinosinusitis After Functional Endoscopic Sinus Surgery (FESS)
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: 082012
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-12

CONDITIONS: Condition of Patient 3 Years After FESS-operation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rhinosinusitis patients: patients having undergone endoscopic sinus surgery (ESS) for bilateral inflammatory sinonasal disease from January 2008 until December 2010.

SUMMARY:
State-of-the-art documents like ARIA and european position paper on rhinosinusitis (EPOS) provide clinicians with evidence-based treatment algorithms for allergic rhinitis (AR) and chronic rhinosinusitis (CRS) respectively (1)(2) . The currently available medications can alleviate symptoms associated with AR and RS, and most patients with RS benefit from endoscopic sinus surgery (ESS). In real life, a significant percentage of patients with AR and CRS continue to experience bothersome symptoms despite adequate treatment. This group with so-called severe chronic upper airway disease (SCUAD) represents a therapeutic challenge (3).

ELIGIBILITY:
Inclusion Criteria:

1. Patients that have undergone bilateral ESS for inflammatory sinonasal disease, without additional sino-nasal surgery after the ESS.
2. Age > 18 and < 75 years.
3. Written informed consent
4. Dutch, French or English speaking patients

Exclusion Criteria:

1. Unilateral ESS
2. Benign and malignant tumor disease
3. Patient with a psychiatric, addictive, or any disorder of which the investigators feel at the time of evaluation for participation in the study that this may compromise the ability to give truly informed consent for participation in this study or provide reliable information on the questionnaire
4. Lack of knowledge of Dutch, French or English

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rhinosinusitis patients
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, MD, Principal Investigator — UZ Leuven
Locations (2):
- Belgium (2):
  - UZ Leuven ORL, Leuven, Vlaams Brabant
  - UZ Leuven, Leuven, Vlaams-Brabant

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rhinosinusitis Patients
Started | 389
Completed | 389
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rhinosinusitis Patients
Number analyzed (Participants) | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 389
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 206
Region of Enrollment [Number; unit: participants]
  Belgium | 389

OUTCOME MEASURES:

1. Primary Outcome: Control Status of Patients With Rhinosinusitis
Description: 1. Percentage of patients with rhinosinusitis that are fully controlled, partly controlled and uncontrolled according to the new european position paper on rhinosinusitis (EPOS) definitions at a mean interval of 3 years after endoscopic sinus surgery.
Time Frame: 3 years after FESS
Measure: Number; unit: percentage of participants
Groups:
- Rhinosinusitis Patients and Status: patients having undergone endoscopic sinus surgery (ESS) for bilateral inflammatory sinonasal disease from January 2008 until December 2010.
Arm/Group | Rhinosinusitis Patients and Status
Number analyzed (Participants) | 389
percentage of participants
  fully controlled three years after ESS | 19.5
  partially controlled three years after ESS | 36.8
  uncontrolled three years after ESS | 43.7

2. Secondary Outcome: Control Nasal Endoscopy
Description: Evaluating of difference in control if nasal endoscopy is performed three years after ESS.
Time Frame: 3 years after ESS
Population: fully controlled status with endoscopic evaluation
Measure: Number; unit: percentage of participants
Arm/Group | Rhinosinusitis Patients
Number analyzed (Participants) | 81
percentage of participants
  fully controlled status with endoscopic evaluation | 8.6
  partially controlled status with endoscopy | 24.7
  uncontrolled status wih endoscopic evaluation | 66.7

3. Other Pre Specified Outcome: Visual Analogue Scale (VAS), Sinonasal Outcome Test (SNOT22) and Short Form (36) Health Survey (SF36) Score Three Years After ESS in Controlled, Partially Controlled and Uncontrolled Group
Description: VAS scores: a measurement of patient's subjective evaluation by indicating a position on a line between two endpoints. Patients will score eight individual symptoms on a scale from 0 until 10, being 0 no trouble and 10 maximum trouble. Finally a mean symptom score will be calculated per symptom.
  The SNOT-22 questionnaire is a validated 22 item questionnaire. patients indicate how much they are affected in eight different areas and identify the 5 most important items. The SNOT-22 total score can range from 0 to 110, with higher scores representing worse quality of life.
  Perceived health status can be evaluated by the 36-item short-form (SF-36). It consists of 36 items covering eight domains. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Time Frame: three years after ESS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rhinosinusitis Patients
Number analyzed (Participants) | 389
units on a scale
  VAS score controlled group | 9.6 (7.9)
  SNOT 22 score controlled group | 10.2 (9.7)
  SF36 score controlled group | 82.1 (14.3)
  VAS score partially controlled group | 22.8 (12)
  SNOT22 score partially controlled group | 21.6 (12.4)
  SF36 score partially controlled group | 76.5 (16.8)
  VAS score uncontrolled group | 45.2 (19.0)
  SNOT22 score uncontrolled group | 43.4 (19.9)
  SF36 score uncontrolled group | 61.9 (19.6)

ADVERSE EVENTS:
Arm/Group | Rhinosinusitis Patients
Serious Adverse Events (participants affected / at risk) | 0/389
Other Adverse Events (participants affected / at risk) | 0/389

LIMITATIONS AND CAVEATS:
patients had to fill in the questionnaire at home, with no help of an expert

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes